CLINICAL TRIAL: NCT06282510
Title: Impact of Nasal Antisepsis on Candida Auris Colonization
Brief Title: Nasal Antisepsis for C. Auris Prevention
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Mary K Hayden (Other)
Collaborators: Rush University Medical Center (Other); RML Specialty Hospital (Other)
Responsible Party: Sponsor-Investigator, Mary K Hayden, Principal Investigator, Rush University Medical Center
Organization: Rush University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 23053003
Record Dates: First submitted 2024-02-08; First posted 2024-02-28 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Candida Auris Infection; Colonization, Asymptomatic
Keywords: Candida auris; Decolonization; Colonization; Infection Prevention; Povidone Iodine; Long-term Care
MeSH Terms: conditions — Candida auris infection; Asymptomatic Infections | interventions — Povidone-Iodine; Iodophors

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intranasal Povidone Iodine (Active Comparator): Nasal iodophor applied twice daily for five days.
  Interventions: Drug: Povidone Iodine Topical
- Control (No Intervention): Routine care.

INTERVENTIONS:
Drug: Povidone Iodine Topical — Topical intranasal povidone iodine (10%) twice daily for 5 days
  Other Names: Iodophor; Betadine; Profend Nasal Decolonization Kit (SKU # X12048)
  Arms: Intranasal Povidone Iodine

SUMMARY:
This is a randomized, controlled, open-label trial of effect of 10% povidone iodine intranasal antisepsis on the detection of Candida auris.

DETAILED DESCRIPTION:
The investigators will assess the effect of nasal antisepsis with 10% povidone iodine on nasal and skin colonization and environmental contamination with C. auris. This topical, widely used antiseptic agent is available over the counter in the U.S. It was chosen for its excellent safety profile, history as a nasal antiseptic for Staphylococcus aureus decolonization, proven in vitro activity against C. auris and feasibility in acute care and nursing home populations. This study will be conducted at 2 long-term acute care hospitals and one acute care hospital in the Chicago, IL region. Participants will first undergo intranasal screening for current C. auris colonization. Participants who grow C. auris from an anterior nares sample will be assigned 1:1 at random to receive intranasal povidone iodine (10% povidone iodine twice daily for up to 5 days) or control (no intranasal treatment). The investigators will perform all study visits during the participants' hospitalization at a participating facility. Samples will be collected on 5 days during the intervention week, then once weekly thereafter. Participants may participate for up to 8 study visits after randomization or until facility discharge, whichever occurs sooner.

ELIGIBILITY:
Inclusion Criteria:

* History of C. auris colonization or infection
* Patient in a participating facility

Exclusion Criteria:

* History of severe allergy to iodine-based products, defined as anaphylaxis or rash
* Currently breastfeeding or pregnant
* Non-English language speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-01-29 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Detection of C. auris from the anterior nares | Through study completion and data analysis in three years (2028)
  Culture detection of C. auris from anterior nares on intervention day 5.

SECONDARY OUTCOMES:
Detection of C. auris from body sites other than anterior nares | Through study completion and data analysis in three years (2028)
  Culture detection of C. auris from body sites other than anterior nares. The investigators will compare detection of C. auris by culture during intervention vs post-intervention periods.
Detection of C. auris from environmental surfaces | Through study completion and data analysis in three years (2028)
  Culture detection of C. auris from participant environmental room surfaces. The investigators will compare detection of C. auris by culture during intervention vs post-intervention periods.
Detection of methicillin-resistant Staphylococcus aureus (MRSA) from body sites other than anterior nares | Through study completion and data analysis in three years (2028)
  Culture detection of MRSA from body sites other than anterior nares. The investigators will compare detection of MRSA by culture during intervention vs post-intervention periods.
Detection of MRSA from environmental surfaces | Through study completion and data analysis in three years (2028)
  Culture detection of MRSA from participant environmental room surfaces. The investigators will compare detection of MRSA by culture during intervention vs post-intervention periods.

OTHER OUTCOMES:
Non-susceptibility of C. auris to povidone iodine | Through study completion and data analysis in three years (2028)
  To assess for development of non-susceptibility of C. auris to povidone iodine, we will evaluate for a ≥4-fold increase in minimal inhibitory concentration (MIC) of povidone iodine pre- and post-intervention
Change in microbiome community | Through study completion and data analysis in three years (2028)
  To assess for microbiome changes during the intervention, anterior nares samples will be analyzed using amplicon and/or metagenomic sequencing approaches. The investigators will compare the microbial community during intervention vs post-intervention periods.

CONTACTS AND LOCATIONS:
Overall Officials: Mary K. Hayden, MD, Principal Investigator — Rush University Medical Center
Locations (3):
- United States (3):
  - Rush University Medical Center, Chicago, Illinois
  - RML Specialty Hospital, Chicago, Illinois
  - RML Specialty Hospital, Hinsdale, Illinois

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-01-13): https://cdn.clinicaltrials.gov/large-docs/10/NCT06282510/ICF_000.pdf